CLINICAL TRIAL: NCT06488326
Title: Effect of Mulberry Leaf Extract Capsule on Blood Glucose Control in Healthy Volunteers
Brief Title: Mulberry Leaf Extract Capsule on Blood Glucose Control in Healthy Volunteers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Mae Fah Luang University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: EC23188-20
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Health, Subjective

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mulberry leaf extract 6 mg capsule (Experimental): Take one capsule of the sample one time.
  Interventions: Drug: Mulberry leaf extract 6 mg capsule
- Mulberry leaf extract 12 mg capsule (Experimental): Take one capsule of the sample one time.
  Interventions: Drug: Mulberry leaf extract 12 mg capsule
- Mulberry leaf extract 18 mg capsule (Experimental): Take one capsule of the sample one time.
  Interventions: Drug: Mulberry leaf extract 18 mg capsule
- Placebo capsule (Placebo Comparator): Take one capsule of the sample one time.
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: Mulberry leaf extract 6 mg capsule — Take one capsule of the sample one time.
  Arms: Mulberry leaf extract 6 mg capsule
Drug: Mulberry leaf extract 12 mg capsule — Take one capsule of the sample one time.
  Arms: Mulberry leaf extract 12 mg capsule
Drug: Mulberry leaf extract 18 mg capsule — Take one capsule of the sample one time.
  Arms: Mulberry leaf extract 18 mg capsule
Drug: Placebo capsule — Take one capsule of the sample one time.
  Arms: Placebo capsule

SUMMARY:
Volunteers will be divided into 4 groups which are mulberry leaf extract 6 mg capsule, mulberry leaf extract 12 mg capsule, mulberry leaf extract 18 mg capsule, and placebo capsule group. They will be tested blood glucose levels (taken from the fingertips) before starting. Then, they will take 1 capsule of the sample one time. After taking the sample for 30 minutes, they will take 50 g of sucrose in 250 ml of water in 5 minutes. Then, they will be tested blood glucose levels (taken from the fingertips) at 30, 60, 90, and 120 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* No diabetes mellitus
* Have blood glucose less than 126 mg/dL
* Wiling to attend the study

Exclusion Criteria:

* Take steroids, psychiatric medicine, thiazide diuretic medicine, and beta blocker medicine within 2 weeks before starting of the study
* Take dietary supplement, herbal substance, and weight-loss medicine within 2 weeks before starting of the study
* Uncontrolled diseases
* History of gastrointestinal tract surgery
* Liver and Kidney diseases
* Pregnancy and lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-02-25 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | 120 minutes
  Volunteers will be measured the blood glucose using blood glucose meter and strip (accuchek) before and after taking the sample for 30, 60, 90, and 120 minutes.